CLINICAL TRIAL: NCT02297321
Title: Evaluation of the Safety and Efficacy of the DeScribe™ Laser Tattoo Removal Accessory Device
Brief Title: Evaluation of the Safety and Efficacy of the DeScribe™ Patch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ON Light Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DeScribe-01
Record Dates: First submitted 2014-11-13; First posted 2014-11-21 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Tattoos
Keywords: tattoos; laser; whitening; patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DeScribe patch (Experimental): Comparison of the number of passes achieved using the Describe patch plus laser compared to laser along
  Interventions: Device: Describe patch

INTERVENTIONS:
Device: Describe patch — Application of Describe patch over tattoo for approximately 5 minutes during Q-switched laser treatment

SUMMARY:
This is a prospective study to evaluate the efficacy and safety of an accessory for laser tattoo removal in allowing multiple passes within a single treatment session.

DETAILED DESCRIPTION:
This is a prospective study to evaluate the efficacy and safety of an accessory for laser tattoo removal in allowing multiple passes within a single treatment session. One half of the tattoo will be randomly assigned laser treatment utilizing the Device (the "Device half"); the other half will receive laser treatment without the Device and serve as the control (the "Control half"). Based on statistical analysis sample size calculations, 30 subjects will be enrolled. The tattoo must be no larger than approximately 2 ½" x 6" or 3" x 5" in size, such that ½ of the tattoo can be covered with a single patch. Each subject will receive a single Treatment Session consisting of 5 minutes. Investigators will administer the standard laser treatment to both the Device and Control sites using well-established tattoo-removal treatment parameters for the laser used. Subjects will return for follow up approximately one month post-treatment. The presence of side effects and adverse events will be assessed and recorded for both Device and Control sites immediately after treatment and at the 1-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects presenting with tattoos approximately 2 ½" x 6" or 3" x 5" or smaller in size.
* Fitzpatrick skin type I - III
* Women of childbearing potential using an accepted form of contraception at least 3 months prior to enrollment and during the study period (i.e., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide, or abstinence)
* Subjects who provide written informed consent
* Subjects who agree to all treatment guidelines and follow-up visits

Exclusion Criteria:

* Subjects younger than 18 years of age
* Subjects with traumatic tattoos
* As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in the study
* Subjects who are pregnant or breastfeeding
* Subjects who are tan
* As per the investigator's discretion, subjects with a history of keloid scarring or abnormal wound healing
* Subjects who have used oral retinoids (isotretinoin or acitretin) within 12 months of study entry
* Subjects currently participating or planning to participate in any other clinical trial specifically designed to treat tattoos during the course of this study and for the duration of their participation in the study
* Subjects who refuse to sign this informed consent form and/or refuse to comply with all study requirements.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of passes with Describe patch | 5 minutes
  Number of passes with Describe patch compared to laser only

SECONDARY OUTCOMES:
Safety assessment: Overall rate and severity of all reported adverse events | immediate post treatment, 1-month post tx
  Overall rate and severity of all reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Brian Biesman, MD, Principal Investigator — Nashville Centre for Laser and Facial Surgery
Locations (1):
- Nashville Centre for Laser and Facial Surgery, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No